CLINICAL TRIAL: NCT03972761
Title: Evaluation of Brain Plasticity in Premature Infants at School Age After Cognitive
Brief Title: Evaluation of Brain Plasticity in Premature Infants at School Age After Cognitive Remediation
Acronym: EPIREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-07; 2019-A00829-48 (Other: ID RCB); RCAPHM19_0023 (Other: Secondary AP-HM number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Premature Childbirth
MeSH Terms: conditions — Premature Birth | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group exposed to cognitive remediation (Active Comparator): Computerized cognitive remediation program. Program performed during inclusion in the EPIREMED patient study (Clinical trial number NCT02757794)
  Interventions: Device: Magnetic Resonance Imaging (MRI) 3 tesla
- Group not exposed to cognitive remediation (Placebo Comparator): Standard remediation performed during inclusion in the EPIREMED patient study (Clinical trial number NCT02757794)
  Interventions: Device: Magnetic Resonance Imaging (MRI) 3 tesla

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) 3 tesla — Functional neuroimaging objectifies the activation of specific areas of the brain

SUMMARY:
Infantile brain plasticity is still a poorly known phenomenon. However, neuropsychological disorders and behavioral deficits are common disorders that can have serious consequences for school enrollment, family and social adjustment, as well as repercussions on future adult lives.

In addition, generally very premature infants (TGP) have identifiable executive function disorders (EF), particularly those involving attentional processes such as working memory (WM).

The main objective of the study is to evaluate the effects of cognitive remediation (CR) strategies on the brain plasticity of the cortical areas involved in the management of WM in school-aged TGP children (8 years).

The secondary objective of the study is to evaluate the action of CR on the development of cortical areas concerned

It is a monocentric, prospective and comparative study of the exposed type (to cognitive remediation) - unexposed. Recruitment and data collection are carried out prospectively, in connection with the original study (EPIREMED). Included patients will be explored by Magnetic Resonance Imaging (MRI) 3 resting state Tesla.

The main hypothesis is that CR strategies have a beneficial effect on the cognitive processing of visual-spatial executive functions, but also on the cortical areas involved in brain plasticity in general (indirect benefits); not to mention the psychological benefits ad hoc to such studies (self-esteem, increased concentration, new stress management strategies put in place).

The ultimate objective of this study is to better understand the mechanisms of cerebral plasticity concerning higher executive functions. Moreover, this study should make it possible to confirm the improvement of the overall fate of the child by better understanding the neuropsychological and anatomical origins of his disorders. Interventions taking into account the environment of the very premature baby are necessary because it is closely linked to the developmental future.

ELIGIBILITY:
Inclusion Criteria:

* Children born between 24 and 34 weeks of amenorrhea and living in the Provence region
* Possessing an intelligence quotient (IQ) greater than 70

Exclusion Criteria:

* Child not understanding French
* Child who did not have all the interventions in the EPIREMED study

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-09-27 (Estimated); Primary Completion 2021-09-26 (Estimated); Study Completion 2021-09-26 (Estimated)

PRIMARY OUTCOMES:
Activation of cortical areas | 24 months
  Hyper activation on the Magnetic Resonance Imaging (MRI) associated with working memory

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No